CLINICAL TRIAL: NCT03531697
Title: A Randomized, Single-blind, Cross-over Study of Loteprednol Etabonate in Adults Undergoing Bilateral Cataract Surgery
Brief Title: Study of Loteprednol Etabonate in Adults Undergoing Bilateral Cataract Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SAN-LE-002
Record Dates: First submitted 2018-04-20; First posted 2018-05-22 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Inflammation Following Ocular Surgery
Keywords: Loteprednol Etabonate
MeSH Terms: interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Generic Loteprednol Etabonate - RLD (Experimental): Period 1: Generic Loteprednol Etabonate - Period 2 (Cross-Over): Reference Listed Drug (RLD)
  Interventions: Drug: Generic Loteprednol Etabonate; Drug: Reference Listed Drug (RLD)
- RLD - Generic Loteprednol Etabonate (Active Comparator): Period 1: Reference Listed Drug (RLD) - Period 2 (Cross-Over): Generic Loteprednol Etabonate
  Interventions: Drug: Generic Loteprednol Etabonate; Drug: Reference Listed Drug (RLD)

INTERVENTIONS:
Drug: Generic Loteprednol Etabonate — Drug
Drug: Reference Listed Drug (RLD) — Drug
  Other Names: Loteprednol Etabonate

SUMMARY:
This study will assess the bioequivalence of Loteprednol Etabonate and the reference listed drug (RLD)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a need for cataract surgery in both eyes and can be dosed in the surgical eyes.
* Non-pregnant, non-lactating females, or women who are post-menopausal (defined as at least 12 months natural, spontaneous amenorrhea), or are naturally or surgically sterile (hysterectomy; bilateral oophorectomy; bilateral tubal ligation with surgery at least 6 weeks prior to study initiation). Females of childbearing potential must have a confirmed absence of pregnancy according to a negative urine pregnancy test and must be using one of the following acceptable birth control methods: Intrauterine device in place for at least 90 days. Barrier method (condom or diaphragm) with spermicide. Stable hormonal contraceptive for at least 90 days prior to study and through study completion. Abstinence (if the subject becomes sexually active during the study she must agree to use the barrier method of birth control [condom or diaphragm and spermicide] for the duration of the study).
* Male subjects should use medically reliable contraception methods such as condom or vasectomy.
* Subjects are able to perform the activities required by the study protocol and have provided written informed consent.

Exclusion Criteria:

* Subjects having an IOP less than 5 mmHg or greater than 24 mmHg.
* Known or suspected allergy or hypersensitivity to loteprednol etabonate or any ingredient in the formulation or container, or to other corticosteroids, including an increase in IOP after steroid instillation.
* Subjects unable to tolerate instillation of study product by the investigator or qualified staff.
* Use of other investigational drugs within 30 days prior to dosing and for the duration of the study.
* Subject has used any medication, by any route, containing loteprednol etabonate within 7 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) assessed by Area Under the Curve (AUC) | upon study completion, up to 1 year
  PK for loteprednol etabonate concentrations in aqueous humor. Area under the concentration versus time curve.
Pharmacokinetic (PK) assessed by rate of drug absorption (Cmax) | upon study completion, up to 1 year
  PK for loteprednol etabonate concentrations in aqueous humor. Maximum observed mean concentration in aqueous humor over the time span specified.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (1):
- Sandoz Investigative Site, Multiple Locations, Canada

IPD SHARING:
Plan to Share IPD: No